CLINICAL TRIAL: NCT01647399
Title: AsthMaP 2: Vitamin D, Steroids, and Asthma in African American Youth
Brief Title: Vitamin D, Steroids, and Asthma in African American Youth
Acronym: AsthMaP2
Status: Completed | Type: Observational
Sponsor: Robert J. Freishtat (Other)
Responsible Party: Sponsor-Investigator, Robert J. Freishtat, Attending Physician, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: R01MD007075-01 (NIH)
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Asthma; Allergy
Keywords: Obesity; Asthma; Vitamin D; Allergy; Genetic; Childhood; Pediatric; cohort; observational; prospective; molecular
MeSH Terms: conditions — Asthma; Hypersensitivity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Phenotypic Clusters: 500 urban youth

SUMMARY:
Asthma has become considerably more prevalent and severe in the U.S. during the last 40 years, particularly affecting youth in urban areas, yet the reasons for this are not clear. There is increasing evidence that vitamin D insufficiency contributes to more severe asthma through increased risk of respiratory infections and decreased sensitivity to glucocorticoids. Indeed, low vitamin D levels are linked with the need for exogenous glucocorticoids and increased asthma severity. Particularly relevant to health disparities, we showed a strong association between vitamin D insufficiency and asthma in urban African American (AA) youth. Importantly, AA youth in ours and other studies had lower vitamin D levels than non-AA participants.

Because AA youth residing in urban Washington, DC have markedly worse asthma than other racial/ethnic groups (e.g. prevalence rate 20% higher than the national rate 15 and emergency department utilization rates up to 5 times the national rates and nearly 10 times the Healthy People 2010 target rate), we will utilize our access to this population at the extreme of asthma disparities to examine the contribution of vitamin D to disparities in the chronic control and acute severity of asthma. The overall goal of this study is to provide critical epidemiological/molecular information that will inform the interpretation of ongoing and impending randomized clinical trials of vitamin D supplementation in asthma, especially with regard to urban AA youth with asthma. We hypothesize that low serum 25-hydroxyvitamin D [25(OH)D] levels are associated with poor chronic asthma control, worse acute asthma severity, and glucocorticoid insensitivity. The knowledge generated by the experiments in this application will be crucial to translation of this inexpensive, easily-accessible, and thereby potentially disparity-reducing prospective therapy for asthma.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 and 20 years of age
* Physician-diagnosed asthma for 1 year or more
* Caretaker/Independent participant willing to sign the written Informed Consent, Assent form when appropriate

Exclusion Criteria:

* Significant, chronic medical illnesses other than asthma
* No access to a phone

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: AshMaP 2 subjects will be enrolled from all the sites in the Children's National Medical Center city-wide pediatric and adolescent health systems sites, including primary care offices (community and hospital-based), specialty clinics, Emergency Departments, and inpatient units.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2012-07; Primary Completion 2017-08 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Serum 25(OH)D measurement by liquid chromatography-tandem mass spectrometry | one year

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Freishtat, MD, MPH, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Maltz L, Matz EL, Gordish-Dressman H, Pillai DK, Teach SJ, Camargo CA Jr, Hubal MJ, Behniwal S, Prosper GD, Certner N, Marwah R, Mansell DM, Nwachukwu F, Lazaroff R, Tsegaye Y, Freishtat RJ. Sex differences in the association between neck circumference and asthma. Pediatr Pulmonol. 2016 Sep;51(9):893-900. doi: 10.1002/ppul.23381. Epub 2016 Jan 15. PMID 26774073
- See also: Related Info — http://www.ChildrensNational.org